CLINICAL TRIAL: NCT01185964
Title: A Phase 1b/2, With Phase 2 Randomized, Study Evaluating the Efficacy of Doxorubicin With or Without a Human Anti-PDGFRα Monoclonal Antibody (IMC-3G3) in the Treatment of Advanced Soft Tissue Sarcoma
Brief Title: A Study of Olaratumab in Soft Tissue Sarcoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14055; I5B-IE-JGDG (Other: Eli Lilly and Company); CP15-0806 (Other: ImClone Systems)
Record Dates: First submitted 2010-08-19; First posted 2010-08-20 (Estimated); Results first posted 2017-04-14 (Actual); Last update posted 2017-04-14 (Actual); Status verified 2017-03

CONDITIONS: Sarcoma, Soft Tissue
Keywords: Sarcoma, Soft Tissue; Advanced Soft Tissue Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — olaratumab; Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Phase 1b: Olaratumab + doxorubicin (Experimental): All cycles are 21 days.
  Cycles 1-8: Olaratumab 15 mg/kg on days 1+8, and doxorubicin 75 mg/m2 on day 1
  All subsequent cycles until progression: Olaratumab 15 mg/kg on days 1+8
  Interventions: Biological: Olaratumab; Drug: doxorubicin
- Phase 2: Olaratumab and doxorubicin (Experimental): All cycles are 21 days.
  Cycles 1-8: Olaratumab 15 mg/kg on days 1+8, and doxorubicin 75 mg/m2 on day 1
  All subsequent cycles until progression: Olaratumab 15 mg/kg on days 1+8
  Interventions: Biological: Olaratumab; Drug: doxorubicin
- Phase 2: Doxorubicin: Optional Olaratumab After Progression (Active Comparator): All cycles are 21 days.
  Cycles 1-8: doxorubicin 75 mg/m2 on day 1 until disease progression.
  At disease progression: optional Olaratumab 15 mg/kg on days 1+8 until further progression.
  Interventions: Drug: doxorubicin

INTERVENTIONS:
Biological: Olaratumab — Olaratumab 15 mg/kg by intravenous transfusion (I.V.) on days 1+8 of a 21-day cycle
  Other Names: LY3012207; IMC-3G3
  Arms: Phase 1b: Olaratumab + doxorubicin; Phase 2: Olaratumab and doxorubicin
Drug: doxorubicin — Doxorubicin 75 mg/m2 by intravenous injection on day 1 of the 21-day cycle.

SUMMARY:
The main purpose of this study is to gather information about the use of an investigational drug called olaratumab with a drug for soft tissue sarcoma called doxorubicin.

ELIGIBILITY:
Inclusion Criteria:

* The participant has histologically- or cytologically-confirmed malignant soft tissue sarcoma
* The participant has advanced soft tissue sarcoma (STS), not amenable to treatment with surgery or radiotherapy
* The participant's Eastern Cooperative Oncology Group (ECOG) performance status is 0-2
* The participant has available tumor tissue from either the primary or metastatic tumor for determination of PDGFRα expression
* The participant has adequate hematologic function as defined by an absolute neutrophil count (ANC) ≥ 1500 μL, hemoglobin ≥ 9.0 g/dL, and a platelet count of 100,000/μL obtained within 2 weeks prior to study entry
* The participant has adequate hepatic function as defined by a total bilirubin ≤ 1.5 mg/dL, and aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 3.0 times the upper limit of normal (ULN)
* The participant has adequate renal function as defined by serum creatinine ≤ 1.5 × the institutional ULN. If creatinine is above the ULN, the participant's creatinine clearance is ≥ 45 mL/min
* Because the teratogenicity of Olaratumab is not known, women of childbearing potential (WOCBP) and sexually active males must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation

Exclusion Criteria:

* The participant has histologically- or cytologically-confirmed Kaposi's sarcoma
* The participant has untreated central nervous system metastases
* The participant received prior treatment with doxorubicin, daunorubicin, idarubicin, and/or other anthracyclines and anthracenediones (ie, mitoxantrone)
* The participant received prior radiation therapy to the mediastinal/pericardial area
* The participant has a history of another primary cancer, with the exception of a) curatively resected nonmelanomatous skin cancer; b) curatively treated cervical carcinoma in situ; or c) other primary solid tumor treated with curative intent, no known active disease present, and no treatment administered during the last 3 years prior to study entry
* The participant is receiving concurrent treatment with other anticancer therapy, including other chemotherapy, immunotherapy, hormonal therapy, radiotherapy, chemo-embolization, targeted therapy, or an investigational agent
* The participant has an elective or a planned major surgery to be performed during the course of the study
* The participant has an uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, requiring parenteral antibiotics, symptomatic congestive heart failure, severe myocardial insufficiency, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* The participant has unstable angina pectoris, angioplasty, cardiac stenting, or myocardial infarction 6 months prior to study entry
* The participant has known immunodeficiency virus (HIV) infection
* The participant, if female, is pregnant or lactating
* The participant has a known allergy to any of the treatment components

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2010-10; Primary Completion 2014-08 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (17):
- United States (17):
  - ImClone Investigational Site, Tucson, Arizona
  - ImClone Investigational Site, Los Angeles, California
  - ImClone Investigational Site, Aurora, Colorado
  - ImClone Investigational Site, Gainesville, Florida
  - ImClone Investigational Site, Orlando, Florida
  - ImClone Investigational Site, Atlanta, Georgia
  - ImClone Investigational Site, Chicago, Illinois
  - ImClone Investigational Site, Rochester, Minnesota
  - ImClone Investigational Site, St Louis, Missouri
  - ImClone Investigational Site, New York, New York
  - ImClone Investigational Site, Charlotte, North Carolina
  - ImClone Investigational Site, Cleveland, Ohio
  - ImClone Investigational Site, Charleston, South Carolina
  - ImClone Investigational Site, Memphis, Tennessee
  - ImClone Investigational Site, San Antonio, Texas
  - ImClone Investigational Site, Seattle, Washington
  - ImClone Investigational Site, Madison, Wisconsin

REFERENCES:
- [Derived] Tap WD, Jones RL, Van Tine BA, Chmielowski B, Elias AD, Adkins D, Agulnik M, Cooney MM, Livingston MB, Pennock G, Hameed MR, Shah GD, Qin A, Shahir A, Cronier DM, Ilaria R Jr, Conti I, Cosaert J, Schwartz GK. Olaratumab and doxorubicin versus doxorubicin alone for treatment of soft-tissue sarcoma: an open-label phase 1b and randomised phase 2 trial. Lancet. 2016 Jul 30;388(10043):488-97. doi: 10.1016/S0140-6736(16)30587-6. Epub 2016 Jun 9. PMID 27291997

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants who had evidence of progressive disease (PD), died, or received optional olaratumab treatment on the doxorubicin (dox) monotherapy arm were considered to have completed the study. This includes participants who discontinued treatment due to non-PD reasons, but had PD at End of Study.
Groups:
- Phase 1b: Olaratumab + Doxorubicin: All cycles are 21 days.
  Cycles 1-8: Olaratumab 15 milligram/kilogram (mg/kg) on days 1+8, and doxorubicin 75 milligram/square meter (mg/m2) on day 1
  All subsequent cycles until progression:
  Olaratumab 15 mg/kg by intravenous IV on days 1+8 of a 21-day cycle
- Phase 2: Olaratumab + Doxorubicin: All cycles are 21 days.
  Cycles 1-8: Olaratumab 15 mg/kg on days 1+8, and doxorubicin 75 mg/m2 on day 1
  All subsequent cycles until progression:
  Olaratumab 15 mg/kg by IV on days 1+8 of a 21-day cycle
- Phase 2: Doxorubicin: All cycles are 21 days.
  Cycles 1-8: doxorubicin 75 mg/m2 on day 1
  At disease progression: optional Olaratumab 15 mg/kg on days 1+8 until further progression.
- Phase 2: Doxorubicin: Optional Olaratumab After Progression: All subsequent cycles: Participants from doxorubicin monotherapy arm received optional Olaratumab 15 mg/kg on days 1+8 of a 21-day cycle.
Period: Phase 1b and Phase 2
Arm/Group | Phase 1b: Olaratumab + Doxorubicin | Phase 2: Olaratumab + Doxorubicin | Phase 2: Doxorubicin | Phase 2: Doxorubicin: Optional Olaratumab After Progression
Started | 15 | 66 | 67 | 0
Received at Least 1 Dose of Study Drug | 15 | 64 | 65 | 0
Completed | 13 | 56 | 58 | 0
Not Completed | 2 | 10 | 9 | 0
Not completed — Withdrawal by Subject | 1 | 6 | 2 | 0
Not completed — Other Therapy Started | 0 | 3 | 3 | 0
Not completed — Participant was beyond maximum weight | 0 | 0 | 1 | 0
Not completed — Adverse Event | 1 | 0 | 2 | 0
Not completed — Off Treatment but alive and on study | 0 | 1 | 1 | 0
Period: Optional Olaratumab Monotherapy on Dox
Arm/Group | Phase 1b: Olaratumab + Doxorubicin | Phase 2: Olaratumab + Doxorubicin | Phase 2: Doxorubicin | Phase 2: Doxorubicin: Optional Olaratumab After Progression
Started | 0 | 0 | 0 | 30 (Participants with disease progression after treatment received olaratumab.)
Completed | 0 | 0 | 0 | 25
Not Completed | 0 | 0 | 0 | 5
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 2
Not completed — Adverse Event | 0 | 0 | 0 | 1
Not completed — On Study Treatment | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1b: Olaratumab + Doxorubicin | Phase 2: Olaratumab + Doxorubicin | Phase 2: Doxorubicin | Total
Number analyzed (Participants) | 15 | 66 | 67 | 148
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.7 (13.16) | 56.8 (12.53) | 55.3 (12.96) | 56.7 (10.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 40 | 34 | 82
  Male | 7 | 26 | 33 | 66
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 6 | 2 | 9
  Not Hispanic or Latino | 14 | 60 | 64 | 138
  Unknown or Not Reported | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Black or African American | 2 | 6 | 5 | 13
  White | 12 | 55 | 60 | 127
  More than one race | 1 | 2 | 0 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 15 | 66 | 67 | 148

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: PFS is measured from randomization until the first radiographic documentation of progression of disease (PD) as defined by Response Evaluation Criteria in Solid Tumors (RECIST) (version 1.1) or death from any cause. Participants who died without PD was considered to have progressed on the day of death. The following censoring rules applied: If no radiologic assessment at baseline or post baseline, participant was censored at the date of randomization. Participants were censored at the day of their last tumor assessment if no PD and were lost to follow up; If death or PD occurred after 2 or more consecutive missing radiographic visits, censoring occurred at the date of the last adequate radiographic visit. If participant started new treatment before PD, the participant was censored at the date of last tumor assessment prior to new therapy. If treatment was discontinued for reasons other than PD and no further assessment, censoring occurred at last tumor assessment.
Time Frame: Randomization Until the First Radiographic Documentation of Objective Progression (Up to 29 Months)
Population: All randomized participants in Phase 2. Per protocol, phase 1b and optional Olaratumab monotherapy data was exploratory and not collected for this outcome measure. Censored Participants = Phase 2 Olaratumab + Doxorubicin = 11 and Doxorubicin = 19.
Measure: Median (95% Confidence Interval); unit: Month
Groups:
- Phase 2: Olaratumab + Doxorubicin: All cycles are 21 days.
  Cycles 1-8: Olaratumab 15 mg/kg on days 1+8, and doxorubicin 75 mg/m2 on day 1
  All subsequent cycles until progression: Olaratumab 15 mg/kg on days 1+8
  Olaratumab 15 mg/kg by IV on days 1+8 of a 21-day cycle
  Doxorubicin 75 mg/m2 by IV on day 1 of the 21-day cycle.
Arm/Group | Phase 2: Olaratumab + Doxorubicin | Phase 2: Doxorubicin
Number analyzed (Participants) | 66 | 67
Month | 6.6 [4.1 to 8.3] | 4.1 [2.8 to 5.4]
Statistical Analysis 1: Comparison: Phase 2: Olaratumab + Doxorubicin vs Phase 2: Doxorubicin; Test type: Superiority or Other; p = 0.0615, Log Rank; Hazard Ratio (HR) = 0.672, 95% CI 2-sided [0.442 to 1.021]

2. Primary Outcome: Number of Participants With Treatment Related Adverse Events (TEAE), Adverse Events (AE) or Serious Adverse Events (SAE) for Safety for the Phase 1b Portion of the Study
Description: All Phase 1b participants who experienced at least 1 TEAE in the Phase 1b portion of the study. Adverse Event with missing relationship to study is counted as related. A summary of SAEs and all other non-serious AEs, regardless of causality, is located in the Reported Adverse Event module.
Time Frame: Baseline Up to 30 Months
Population: All participants in Phase 1b.
Measure: Number; unit: participants
Groups:
- Phase 1b: Olaratumab + Doxorubicin: All cycles are 21 days.
  Cycles 1-8: Olaratumab 15 milligram/kilogram (mg/kg) on days 1+8, and doxorubicin 75 milligram/square meter (mg/m2) on day 1
  All subsequent cycles until progression: Olaratumab 15 mg/kg on days 1+8
  Olaratumab 15 mg/kg by intravenous IV on days 1+8 of a 21-day cycle
  Doxorubicin 75 mg/m2 by intravenous injection on day 1 of the 21-day cycle.
Arm/Group | Phase 1b: Olaratumab + Doxorubicin
Number analyzed (Participants) | 15
participants
  Any AE | 14
  Any SAE | 7

3. Secondary Outcome: Number of Participants With AEs and SAEs for Phase 2 Portion
Description: A summary of SAEs and all other non-serious AEs, regardless of causality, is located in the Reported Adverse Event module.
Time Frame: Baseline, Up to 30 Months
Population: All randomized participants who received at least 1 dose of study drug in Phase 2 and optional Olaratumab monotherapy.
Measure: Number; unit: participants
Arm/Group | Phase 2: Olaratumab + Doxorubicin | Phase 2: Doxorubicin | Phase 2: Doxorubicin: Optional Olaratumab After Progression
Number analyzed (Participants) | 64 | 65 | 30
participants
  Any AE | 63 | 64 | 24
  Any SAE | 27 | 26 | 9

4. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the date of randomization to the date of death from any cause. Reasons for censoring OS were that participant was known to be alive, participant was lost to follow up during the study or participant withdrew consent to follow up.
Time Frame: Randomization to the Date of Death From Any Cause (Up To 47 Months)
Population: All randomized participants in Phase 2. Per protocol, phase 1b and optional Olaratumab monotherapy data was exploratory and not collected for this outcome measure. Censored participants = Phase 2 Olaratumab + Doxorubicin = 27 and Doxorubicin = 15.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 2: Olaratumab + Doxorubicin | Phase 2: Doxorubicin
Number analyzed (Participants) | 66 | 67
Months | 26.5 [20.9 to 31.7] | 14.7 [9.2 to 17.1]
Statistical Analysis 1: Comparison: Phase 2: Olaratumab + Doxorubicin vs Phase 2: Doxorubicin; Test type: Superiority or Other; p = 0.0003, Log Rank; Hazard Ratio (HR) = 0.463, 95% CI 2-sided [0.301 to 0.710]

5. Secondary Outcome: Percentage of Participants With Objective Response (Objective Response Rate)
Description: Objective Response Rate (ORR) is confirmed best overall tumor response of CR or PR. According to RECIST v1.1, PR defined as a >30% decrease in the sum of the longest diameters (LD) of the target lesions, taking as reference the baseline sum of the LD; CR was defined as the disappearance of all target and non-target lesions. Percentage of participants was calculated as: total number of participants with a best tumor response of PR or CR among participants counted in the denominator/total number of participants treated with any amount of study drug, who has a complete radiographic assessment at baseline, and who has at least 1 complete radiographic assessment at postbaseline x 100%.
Time Frame: Randomization Until Progressive Disease (Up to 30 Months)
Population: All randomized participants in Phase 2 and optional Olaratumab monotherapy.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2: Olaratumab + Doxorubicin | Phase 2: Doxorubicin | Phase 2: Doxorubicin: Optional Olaratumab After Progression
Number analyzed (Participants) | 66 | 67 | 30
percentage of participants | 18.2 [9.8 to 29.6] | 11.9 [5.3 to 22.2] | 0 [0.0 to 11.6]

6. Secondary Outcome: Percentage of Participants Who Are Progression-Free (PFS) at 3 Months
Description: (PFS) rate is defined as the percentage of participants that are alive and progression-free 3 months after randomization. PFS is measured from randomization until the first radiographic progressive disease as defined by RECIST (version 1.1) or death from any cause. Participants who died without PD were considered to have progressed on the day of death. Censoring applied: If no radiologic assessment at baseline or post baseline, participant was censored at the date of randomization or the day of their last tumor assessment if no PD and were lost to follow up; If death or PD occurred after 2 or more consecutive missing radiographic visits, censoring occurred at the date of the last radiographic visit. If participant started new treatment before PD, participant was censored at the date of last tumor assessment prior to new therapy. If treatment was discontinued for reasons other than PD and no further assessment, censoring occurred at last tumor assessment.
Time Frame: Randomization Until First Radiographic PD or Death from Any Cause (Up to 3 Months)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2: Olaratumab + Doxorubicin | Phase 2: Doxorubicin
Number analyzed (Participants) | 66 | 67
percentage of participants | 69.0 [55.7 to 78.9] | 59.9 [45.9 to 71.4]

7. Secondary Outcome: Pharmacokinetic (PK) Maximum Concentration (Cmax) Cycle 1 Day 1, Cycle 3 Day 1 of Olaratumab
Time Frame: Cycle 1 Day 1: Preinfusion, End of Infusion,1hr,48hr,72hr,168 hr Post infusion; Cycle 3 Day 1:Preinfusion, End of Infusion,1hr,24hr,48hr,72hr,168hr Post Infusion
Population: All participants who had evaluable PK data in Phase 1b and Phase 2. Per protocol, optional Olaratumab monotherapy data was exploratory and not collected for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram/milliliter (μg/mL )
Groups:
- Phase 1b and Phase 2 Olaratumab + Doxorubicin: All cycles are 21 days.
  Cycles 1-8: Olaratumab 15 milligram/kilogram (mg/kg) on days 1+8, and doxorubicin 75 milligram/square meter (mg/m2) on day 1
  All subsequent cycles until progression:
  Olaratumab 15 mg/kg by intravenous IV on days 1+8 of a 21-day cycle
Arm/Group | Phase 1b and Phase 2 Olaratumab + Doxorubicin
Number analyzed (Participants) | 60
nanogram/milliliter (μg/mL )
  Cycle 1 Day 1 (n=60) | 284 (23.3)
  Cycle 3 Day 1 (n=30) | 404 (31.6)

8. Secondary Outcome: PK: Minimum Concentration (Cmin) Cycle 1 Day 8, Cycle 3 Day 8 of Olaratumab
Time Frame: Cycle 1 Day 8: Preinfusion, 1hr,72hr,168hr Post Infusion; Cycle 3 Day 8: Preinfusion,1hr, 24hr,72hr,168hr Post Infusion
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Groups:
- Phase 1b and Phase 2: Olaratumab + Doxorubicin: All cycles are 21 days.
  Cycles 1-8: Olaratumab 15 milligram/kilogram (mg/kg) on days 1+8, and doxorubicin 75 milligram/square meter (mg/m2) on day 1
  All subsequent cycles until progression:
  Olaratumab 15 mg/kg by intravenous IV on days 1+8 of a 21-day cycle
Arm/Group | Phase 1b and Phase 2: Olaratumab + Doxorubicin
Number analyzed (Participants) | 52
μg/mL
  Cycle 1 Day 8 (n=52) | 66.5 (40.4)
  Cycle 3 Day 8 (n=29) | 123 (39.6)

9. Secondary Outcome: PK: Area Under Concentration Curve Versus Time (AUCτ) Cycle 1 Day 8, Cycle 3 Day 8 of Olaratumab
Description: AUCτ = area under the concentration versus time curve during one dosing interval with a measurable concentration.
Time Frame: Cycle 1 Day 8:Preinfusion,1hr,72hr,168hr Post Infusion; Cycle 3 Day 8: Preinfusion,1hr,24hr,72hr,168hr Post Infusion
Population: All participants who had evaluable PK data in Phase1b and Phase 2. Per protocol, optional Olaratumab monotherapy data was exploratory and not collected for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram•hour/milliliter (μg•h/mL)
Arm/Group | Phase 1b and Phase 2: Olaratumab + Doxorubicin
Number analyzed (Participants) | 7
microgram•hour/milliliter (μg•h/mL)
  Cycle 1 Day 8 (n=7) | 39200 (29.0)
  Cycle 3 Day 8 (n=4) | 47300 (35.0)

10. Secondary Outcome: PK: Half-Life (T1/2) Cycle 1 Day 8, Cycle 3 Day 8 of Olaratumab
Time Frame: Cycle 1 Day 8:Preinfusion,1hr,72hr,168hr Post Infusion; Cycle 3 Day 8: Preinfusion,1hr,24hr,72hr,168hr Post Infusion
Population: as for outcome 7
Measure: Geometric Mean (Full Range); unit: Days
Arm/Group | Phase 1b and Phase 2: Olaratumab + Doxorubicin
Number analyzed (Participants) | 7
Days
  Cycle 1 Day 8 (n=7) | 6.70 [4.32 to 9.55]
  Cycle 3 Day 8 (n=2) | 9.80 [6.67 to 14.4]

11. Secondary Outcome: Percentage of Participants With Anti-Olaratumab Antibody Assessment
Description: Participants with Treatment Emergent (TE) anti-olaratumab antibodies were participants with a 4-fold increase (2 dilutions) increase over a positive baseline antibody titer or for a negative baseline titer, a participant with an increase from the baseline to a level of 1:20.
Time Frame: Baseline, Up to 30 Months
Population: All participants who had baseline and post baseline anti-olaratumab antibodies.
Measure: Number; unit: percentage of participants
Arm/Group | Phase 1b: Olaratumab + Doxorubicin | Phase 2: Olaratumab + Doxorubicin | Phase 2: Doxorubicin: Optional Olaratumab After Progression
Number analyzed (Participants) | 11 | 58 | 16
percentage of participants | 9.1 | 5.2 | 6.3

ADVERSE EVENTS:
Description: All participants who received at least one dose of study drug.
Arm/Group | Phase 1b: Olaratumab + Doxorubicin | Phase 2: Olaratumab + Doxorubicin | Phase 2: Doxorubicin | Phase 2: Doxorubicin: Optional Olaratumab After Progression
Serious Adverse Events (participants affected / at risk) | 7/15 | 27/64 | 26/65 | 9/30
Other Adverse Events (participants affected / at risk) | 14/15 | 63/64 | 64/65 | 24/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1b: Olaratumab + Doxorubicin (N=15) | Phase 2: Olaratumab + Doxorubicin (N=64) | Phase 2: Doxorubicin (N=65) | Phase 2: Doxorubicin: Optional Olaratumab After Progression (N=30)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (3) | 8 (8) | 8 (9) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 3 (5) | 3 (3) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastric perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (3) | 1 (1) | 2 (2) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (4) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Device breakage (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Disease progression (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Hepatic haemorrhage (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Actinomycotic skin infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutropenic sepsis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Anastomotic ulcer (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wound necrosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Troponin increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 0 (0) | 2 (2)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Phase 1b: Olaratumab + Doxorubicin (N=15) | Phase 2: Olaratumab + Doxorubicin (N=64) | Phase 2: Doxorubicin (N=65) | Phase 2: Doxorubicin: Optional Olaratumab After Progression (N=30)
Anaemia (Blood and lymphatic system disorders) | 11 (42) | 26 (87) | 24 (31) | 5 (12)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 3 (3) | 2 (2)
Leukopenia (Blood and lymphatic system disorders) | 7 (15) | 16 (47) | 5 (11) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 5 (8) | 28 (83) | 13 (18) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 5 (7) | 14 (56) | 10 (14) | 0 (0)
Left ventricular dysfunction (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 2 (2) | 1 (1) | 3 (3) | 2 (2)
Tachycardia (Cardiac disorders) | 1 (1) | 4 (5) | 3 (3) | 1 (1)
Deafness unilateral (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 7 (8) | 2 (2) | 0 (0)
Lacrimation increased (Eye disorders) | 1 (1) | 4 (4) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 6 (6) | 1 (1) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 5 (8) | 5 (5) | 2 (2)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 3 (4) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 8 (10) | 2 (3) | 1 (1)
Anal fissure (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 4 (7) | 21 (38) | 21 (26) | 3 (4)
Diarrhoea (Gastrointestinal disorders) | 4 (5) | 22 (35) | 15 (21) | 5 (7)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 6 (7) | 6 (6) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 6 (6) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (2) | 4 (7) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 4 (5) | 4 (4) | 1 (1)
Nausea (Gastrointestinal disorders) | 8 (12) | 47 (99) | 33 (55) | 6 (7)
Proctalgia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (2) | 1 (2)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 2 (3) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 4 (4) | 11 (13) | 10 (14) | 1 (1)
Vomiting (Gastrointestinal disorders) | 5 (5) | 29 (36) | 12 (16) | 5 (7)
Asthenia (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Catheter site rash (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Chills (General disorders) | 1 (1) | 4 (4) | 2 (2) | 3 (3)
Fatigue (General disorders) | 9 (16) | 44 (83) | 45 (73) | 6 (9)
Mucosal inflammation (General disorders) | 2 (2) | 17 (28) | 12 (28) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 8 (8) | 3 (3) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 10 (14) | 7 (10) | 4 (5)
Pyrexia (General disorders) | 2 (2) | 15 (18) | 12 (17) | 3 (3)
Portal vein thrombosis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 2 (2) | 4 (4) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 8 (8) | 4 (4) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 3 (3) | 3 (3) | 2 (2)
Vaginal infection (Infections and infestations) | 1/8 (1) | 0 (0) | 0 (0) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Incision site complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 2 (2) | 2 (5) | 0 (0) | 1 (1)
Tooth fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound complication (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 3 (5) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 2 (3) | 3 (3) | 1 (1) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Ejection fraction decreased (Investigations) | 1 (1) | 5 (5) | 4 (4) | 0 (0)
International normalised ratio increased (Investigations) | 4 (5) | 2 (2) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 5 (18) | 2 (6) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 12 (25) | 9 (14) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 6 (11) | 3 (3) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 7 (8) | 7 (7) | 2 (2)
White blood cell count decreased (Investigations) | 0 (0) | 12 (46) | 7 (13) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 6 (6) | 19 (22) | 13 (13) | 3 (4)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 6 (6) | 6 (9) | 2 (4)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 4 (10) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 (4) | 4 (4) | 3 (4) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 2 (2) | 5 (5) | 2 (2) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 8 (10) | 5 (9) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 (2) | 5 (6) | 1 (1) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 3 (4) | 6 (6) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 2 (3) | 2 (2) | 2 (5) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 8 (8) | 2 (3) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 10 (17) | 6 (6) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 5 (5) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (2) | 10 (20) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 8 (10) | 1 (2) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (5) | 2 (2) | 1 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 6 (8) | 2 (2) | 1 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 15 (19) | 1 (1) | 2 (2)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2) | 3 (3) | 1 (2)
Dizziness (Nervous system disorders) | 1 (1) | 6 (7) | 10 (12) | 5 (7)
Dysgeusia (Nervous system disorders) | 0 (0) | 6 (7) | 3 (3) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 13 (15) | 6 (7) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 2 (2) | 3 (3) | 1 (1)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 2 (2) | 8 (8) | 5 (5) | 2 (2)
Parosmia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 3 (5) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 3 (3) | 7 (8) | 2 (2) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 4 (4) | 2 (2) | 0 (0)
Hallucination (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 8 (9) | 6 (6) | 2 (2)
Chromaturia (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 4 (4) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0/8 (0) | 3/40 (3) | 0/34 (0) | 0/14 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 14 (16) | 12 (17) | 3 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 11 (14) | 12 (13) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) | 2 (3) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4) | 2 (2) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 12 (15) | 3 (4) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (5) | 2 (2) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 1 (2) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 6 (6) | 33 (41) | 26 (32) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2) | 4 (5) | 4 (4) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | 1 (1) | 0 (0)
Nail discolouration (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | 1 (1) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (1) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 2 (2)
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Embolism (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 4 (4) | 4 (4) | 0 (0)
Jugular vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days